CLINICAL TRIAL: NCT02788903
Title: A Patient-Centered PaTH to Addressing Diabetes: Impact of State Health Policies on Diabetes Outcomes and Disparities and Enhancement Study: Telemedicine Access and Severe Disease Outcomes in Patients With Diabetes and Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Brief Title: A Patient-Centered PaTH to Addressing Diabetes
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jennifer Kraschnewski, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Other Study IDs: PCORI; NEN-1509-32304 (Other Grant/Funding Number: PCORI Contract Number)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Diabetes; Covid19
Keywords: Obesity Counseling; telemedicine
MeSH Terms: conditions — Obesity; Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes: During year 1 of the proposed project, the investigative team will identify a valid cohort of patients with type 2 diabetes using EHR data. The cohort of patients under study will be defined as all patients age 18 and older with an indication of type 2 diabetes during the proposed study time frame (2009-2019).
  Interventions: Other: Weight Counseling
- Pre-Diabetes: The cohort of patients under study will be defined as patients age 18 and older who are at risk for the development of diabetes, based on being overweight. Patients seen at one of the six PaTH institutions will be included in the at-risk cohort if they have a BMI ≥ 25 kg/m2, based on most recent recorded weight and at least one recorded height.
  Interventions: Other: Weight Counseling

INTERVENTIONS:
Other: Weight Counseling — This is a natural experiment which will observe the impact of weight counseling by primary care physicians on patient outcomes.

SUMMARY:
The overarching goal of this proposal is to understand the comparative effectiveness of obesity counseling as covered by CMS in improving weight loss for adults either with or at high risk of type 2 diabetes. CMS and most insurers now include obesity screening and counseling benefits, with no cost sharing to patients. Since overweight patients are at highest risk for diabetes, improved weight management services could prevent diabetes and its negative health outcomes. Beneficiaries with obesity are eligible for up to 20 face-to-face visits for weight counseling in the primary care setting. The investigators propose comparing weight and diabetes outcomes in three states using EHR and claims data before and after this policy was implemented by leveraging the novel infrastructure of the Patient-Centered Outcomes Research Institute-funded PaTH Clinical Data Research Network. Following developments during the COVID-19 pandemic, the investigators further plan to leverage our study infrastructure across five health systems to understand the comparative effectiveness of telemedicine approaches for providing outpatient care for patients with or at risk of type 2 diabetes and how these approaches impact the subgroup of patients with COVID-19.

DETAILED DESCRIPTION:
Aim 1: Evaluate the impact of universal preventive service coverage for obesity screening and counseling on weight loss, diabetes incidence, and diabetes outcomes, in patients with diabetes or at high risk for diabetes (defined by body mass index (BMI) ≥ 25). The investigators will determine how the annual probability of receiving obesity and/or nutritional counseling (as defined by Current Procedural Terminology (CPT) code) changed pre- and post-policy across all insurers in a cohort of patients with diabetes and at high risk for diabetes. The investigators hypothesize that individual patients are more likely to receive counseling following coverage implementation. Further, the investigators hypothesize that patients who receive a greater number of face-to-face visits will have greater weight loss compared to those who receive fewer visits.

Aim 2: Compare patient weight loss and diabetes-related outcomes among those who receive obesity screening and counseling to those who do not, following implementation of preventive service coverage. The investigators will examine post-policy impact of obesity screening and counseling in a cohort of patients with diabetes and at high risk for diabetes. Specific outcomes to be examined include weight loss, diabetes incidence, and diabetes outcomes (including hemoglobin A1c, controlled blood pressure, use of a statin medication). Further, the investigators will determine patient characteristics, including demographics (age, race/ethnicity, rurality), and practice characteristics, including provider type, and their impact on receiving/providing obesity screening and counseling. Understanding patient and practice characteristics most likely to engage in obesity counseling can identify best practices and inform how to increase engagement by both patients and providers.

Aim 3: To understand the impact of telemedicine access (telephonic and/or virtual visits) compared to no telemedicine visits for outpatient care for patients with, or at risk of, type 2 diabetes during the pandemic on patient-centered outcomes including hemoglobin A1c and healthcare utilization, with sub-group analysis of patients with COVID-19;

Aim 4: To evaluate the risk of severe COVID-19 disease (defined by hospitalization and mortality) in patients with diabetes and/or elevated BMI, with a focus on identifying modifiable factors (i.e., medication use, treatment timeline/location, chronic comorbid conditions) and associated with improved outcomes to inform immediate intervention and future study.

ELIGIBILITY:
Inclusion Criteria:

Patients with Diabetes

* Ages 18 and older
* Indication of Type 2 Diabetes as defined using a clinically validated algorithm: type 2 diabetes mellitus on the problem list, diabetes-specific medications, hemoglobin A1c (HbA1c) results > 6.5%, or one inpatient diagnosis code or two out-patient diagnosis codes for type 2 diabetes (ICD-9 codes 250.xx)
* patients who have either: (1) visited a primary care doctor from one of the PaTH health systems in the past 3 years (since January 1, 2012), or (2) for whom claims data are available

Patients with Pre-Diabetes (At risk):

* Ages 18 and older
* BMI > 25 kg/m2
* patients who have either: (1) visited a primary care doctor from one of the PaTH health systems in the past 3 years (since January 1, 2012), or (2) for whom claims data are available

Patients with COVID-19:

* Ages 18 and older
* Patients with a diagnosis of COVID-19

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected through the PaTH Clinical Data Research Network (CDRN), a partnership of six academic health systems (Penn State Hershey Medical Center, University of Pittsburgh Medical Center, Temple Health System, Johns Hopkins Health System, University of Utah and Geisinger Health System) creating an electronic health record (EHR)-based data infrastructure across three states (Maryland, Pennsylvania, and Utah).
Sampling Method: Probability Sample
Enrollment: 2622164 (Actual)
Dates: Start 2016-03; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Kraschnewski, MD, MPH, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center

REFERENCES:
- [Derived] Yeh HC, Kraschnewski JL, Kong L, Lehman EB, Heilbrunn ES, Williams P, Poger JM, Francis E, Bryce CL. Hospitalization and mortality in patients with COVID-19 with or at risk of type 2 diabetes: data from five health systems in Pennsylvania and Maryland. BMJ Open Diabetes Res Care. 2022 Jun;10(3):e002774. doi: 10.1136/bmjdrc-2022-002774. PMID 35680172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants' data was analyzed as part of a secondary data analysis analyzing de-identified EHR and Claims data. Participants did not consent to participate in this study.
Pre-assignment Details: Participants were not randomized for this study.
Groups:
- Diabetes: During year 1 of the proposed project, the investigative team will identify a valid cohort of patients with type 2 diabetes using EHR data. The cohort of patients under study will be defined as all patients age 18 and older with an indication of type 2 diabetes during the proposed study time frame (2009-2019).
  Weight Counseling: This is a natural experiment which will observe the impact of weight counseling by primary care physicians on patient outcomes.
  Telemedicine: This is a natural experiment which will observe the impact of telemedicine approaches for providing outpatient care for patients with or at risk of type 2 diabetes
Period: Overall Study
Arm/Group | Diabetes | Pre-Diabetes
Started | 567908 | 2054256
Completed | 567908 | 2054256
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes | Pre-Diabetes | Total
Number analyzed (Participants) | 567,908 | 2,054,256 | 2622164
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-24 years | 10,371 | 259,691 | 270062
  Age: 25-34 years | 23,169 | 355,885 | 379054
  Age: 35-44 years | 51,885 | 340,065 | 391950
  Age: 45-54 years | 105,646 | 374,446 | 480092
  Age: 55-64 years | 151,061 | 346,075 | 497136
  Age: 65-74 years | 131,104 | 224,386 | 355490
  Age: >75 years | 94,672 | 153,708 | 248380
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 287,725 | 1,167,327 | 1455052
  Sex: Male | 280,170 | 886,884 | 1167054
  Sex: Other/Missing | 13 | 45 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29,211 | 105,438 | 134649
  Not Hispanic or Latino | 514,125 | 1,855,612 | 2369737
  Unknown or Not Reported | 24,572 | 93,206 | 117778
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1,860 | 4,725 | 6585
  Race: Asian | 10,809 | 35,410 | 46219
  Race: Black | 79,732 | 216,860 | 296592
  Race: Native Hawaiin or Other Pacific Islander | 1,311 | 4,413 | 5724
  Race: White | 438,948 | 1,667,767 | 2106715
  Race: Multiple Race | 397 | 1,879 | 2276
  Race: Other/Missing | 34,851 | 123,202 | 158053
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Rural | 31,402 | 92,934 | 124336
  United States: Urban | 470,209 | 1,744,529 | 2214738
  United States: Missing | 66,297 | 216,793 | 283090
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (7.9) | 30.9 (6.2) | 31.55 (7.14)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 75.0 (7.7) | 76.6 (7.4) | 75.24 (10.67)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 130.4 (12.1) | 126.0 (11.9) | 127.03 (17.07)
Hemoglobin A1c [Mean (Inter-Quartile Range); unit: mg/dL] | 7.0 [6.3 to 8.1] | 5.6 [5.3 to 5.8] | 6.9 [6.3 to 8.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Used the Intensive Behavioral Therapy (IBT) Service
Description: Number of patients who utilized IBT services was assessed in both the diabetes and pre-diabetes cohorts using code G0447.
Time Frame: 11 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
Participants | 2417 | 3731

2. Primary Outcome: Change in Weight During Counseling Program
Description: Weight change during counseling and/or % of weight change during program and maintained over remaining time period will be assessed in both the diabetes and pre-diabetes cohorts.
Time Frame: 11 years
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
lbs | 206.8 (55.0) | 194.8 (44.9)

3. Primary Outcome: Hemoglobin A1c
Description: A1c of patients who received a telehealth visit and COVID-19 diagnosis in both the diabetes and pre-diabetes cohorts.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
mmol/mol | 6.6 (1.5) | 6.6 (1.5)

4. Primary Outcome: Number of Participants Diagnosed With COVID-19 Who Were Hospitalized
Description: Number of Participants Diagnosed with COVID-19 Who Were Hospitalized in both the diabetes and pre-diabetes cohorts.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
Participants | 1,025 | 1,379

5. Secondary Outcome: Number of Patients Who Received Telehealth and Were Hospitalized With a COVID-19 Diagnosis
Description: Number of patients who received telehealth and were hospitalized with a COVID-19 diagnosis in both the diabetes and pre-diabetes cohorts.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
Participants | 639 | 838

6. Secondary Outcome: Number of Patients With Uncontrolled Blood Pressure
Description: The number of patients with uncontrolled blood pressure (SBP > 140, DBP > 90 all the time, defined for 1-year prior to first IBTb visit, and 1-year after) in the diabetes and pre-diabetes cohorts
Time Frame: 11 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
Participants | 300,665 | 928,366

7. Secondary Outcome: Number of Patients With Uncontrolled Hemoglobin A1c
Description: The number of patients with uncontrolled hemoglobin A1c (HbA1cc > 9 any time, defined for 1-year prior to first IBTb visit, and 1-year after) in the diabetes and pre-diabetes cohorts.
Time Frame: 11 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
Participants | 79,046 | 164

8. Secondary Outcome: Number of Patients With a COVID-19 Diagnosis and ICU Use, Ventilator Use, or Death
Description: Incidence of ICU admission, ventilator use, or death in patients with a COVID-19 diagnosis in both the diabetes and pre-diabetes cohorts.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes | Pre-Diabetes
Number analyzed (Participants) | 567,908 | 2,054,256
Participants | 586 | 500

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected as patients were not enrolled in the study. This study included only secondary data.
Description: Adverse event data were not collected as patients were not enrolled in the study. This study included only secondary data.
Groups:
- COVID-19: This cohort of patients will be defined as patients age 18 and older who have received a diagnosis of COVID-19.
  Telemedicine: This is a natural experiment which will observe the impact of telemedicine approaches for providing outpatient care for patients with or at risk of type 2 diabetes
Arm/Group | Diabetes | Pre-Diabetes | COVID-19
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT02788903/Prot_SAP_000.pdf